CLINICAL TRIAL: NCT00892580
Title: Biomarker Testing and DNA Collection in Subjects Participating in an Open-Label, Flexible-Dose Evaluation of the Efficacy, Safety, and Tolerability of STX209 in the Treatment of Irritability in Subjects With Autism Spectrum Disorders
Brief Title: Biomarker and DNA Collection in Subjects Participating in Protocol 22003
Status: Completed | Type: Observational
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 22003A
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Fragile X Syndrome
Keywords: fragile X syndrome; biomarkers
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood, plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: STX209 — collection of serum for DNA to elucidate a potential biomarker for patients with ASD

SUMMARY:
The subjects that meet the inclusion and exclusion criteria and consent to participate in protocol 22003 will be offered participation in 22003A which will evaluate secreted protein before and after treatment with STX209 and placebo to determine if they correlate with effectiveness of treatment or susceptibility to treatment with STX209. These same subjects will also be asked to contribute a blood sample for DNA (deoxyribonucleic acid) collection. The investigators will study the DNA to determine if STX209 works better in people with specific gene variations, or to find new gene variations that predict how well STX209 works.

ELIGIBILITY:
Inclusion Criteria:

* The Autism Spectrum Disorder subjects that meet the inclusion and exclusion criteria and consent to participate in protocol 22003

Exclusion Criteria:

* The Autism Spectrum Disorder subjects that meet the inclusion and exclusion criteria and consent to participate in protocol 22003

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Autism Spectrum Disorder subjects
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Biomarker | june 2013
  evaluation of DNA for ASD to elucidate a potential biomaker

CONTACTS AND LOCATIONS:
Overall Officials: Craig Erikson, MD, Principal Investigator — Riley Hospital for Children; Bryan King, MD, PhD, Principal Investigator — Seattle Children's Hospital; James McCracken, MD, Principal Investigator — University of California, Los Angeles; Lawrence Scahill, PhD, Principal Investigator — Yale University; Linmarie Sikich, MD, Principal Investigator — University of North Carolina Neurosciences Hospital; Jeremy Veenstra-VanderWeele, MD, Principal Investigator — Vanderbilt Kennedy Center; Lawrence Ginsberg, MD, Principal Investigator — Red Oaks Psychiatry Associates, PA; Raun Melmed, MD, Principal Investigator — Southwest Autism Research & Resource Center
Locations (8):
- United States (8):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - Yale Child Study Center, New Haven, Connecticut
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of North Carolina Neurosciences Hospital, Chapel Hill, North Carolina
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Red Oaks Psychiatry Associates, PA, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington